CLINICAL TRIAL: NCT05362162
Title: Comparison of Intermediate Cervical Plexus Block and Superficial Cervical Plexus Block for Central Venous Catheterization; Prospective and Randomized Study
Brief Title: Comparison of Intermediate Cervical Plexus Block and Superficial Cervical Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Central Venous Catheterization
Record Dates: First submitted 2022-05-01; First posted 2022-05-05 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-05

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Cervical Plexus Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Active Comparator): Superficial cervical plexus block; After asepsis and antisepsis are achieved, it will be performed by injecting 10 ml of the local anesthetic agent into the subcutaneous area in the anterolateral neck region, from the anatomical region that fits the carotid artery bifurcation point, under the guidance of USG.
  Interventions: Procedure: cervical plexus block
- Group I (Active Comparator): Intermediate cervical plexus block; After asepsis and antisepsis are achieved, it will be performed by injecting 10 ml of the local anesthetic agent under the investing fascia from the anatomical region that fits the carotid artery bifurcation point under the guidance of USG.
  Interventions: Procedure: cervical plexus block

INTERVENTIONS:
Procedure: cervical plexus block — local anesthetic agent injection into the either Superficial or intermediate area

SUMMARY:
Central venous catheterization is a common procedure in hospitals. Internal jugular vein (IJV) cannulation is the most preferred vein for this purpose. During the procedure, infiltration of local anesthetic (LA) agents into the skin and subcutaneous tissues is a commonly used method to provide patient comfort and reduce pain. There is an increasing need to improve the quality of health care delivery. An important component of health service quality is patient satisfaction. The aim of this study is to compare the superficial cervical plexus block and the intermediate cervical plexus block applied under the guidance of ultrasound in terms of patient satisfaction and procedural comfort during central catheterization of the internal jugular vein.

DETAILED DESCRIPTION:
This prospective randomized study will be performed on patients undergoing central venous catheterization into the internal jugular vein. Patients who agreed to participate in the study will be divided into two groups using the closed-envelope randomization method; Group S: Superficial cervical plexus block group Group I: Intermediate cervical plexus group

After routine monitoring and RAMSEY 2 level sedation is achieved, a superficial or intermediate cervical plexus block will be applied according to randomization by a researcher experienced in a peripheral block. Patient pain level (to be evaluated with the Numeric Pain Rating Scale) during the block and catheterization procedure (first needle insertion, dilatation, catheter placement, and suture phase). Thirty minutes after the procedure, patient satisfaction will be evaluated with a Likert-type scale.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteer patients who require central catheterization into the internal jugular vein for any reason
* Patients with mental and health status who can understand the research questions.
* Patients who read the informed consent form and gave a signed declaration of acceptance

Exclusion Criteria:

* Patients with psychiatric disorders
* Patients who are in poor general condition and require urgent intervention
* Patients who cannot answer the survey questions
* Patients followed as intubated
* Patients with hypersensitivity to the local anesthetic agents to be used in the study or to the substances contained in it.
* Patients with contraindications for cervical plexus block application
* Patients who are unwilling to participate in the study for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
patient satisfaction and procedural comfort | 30 minutes following block
  Likert scale; Very satisfied, Satisfied, Neither satisfied nor dissatisfied, Dissatisfied, and Very dissatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Betul Kozanhan, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No